CLINICAL TRIAL: NCT05682378
Title: An Open-label, Single Arm, Multicenter Extension Study to Evaluate Long-term Safety and Tolerability of Inclisiran in Participants With Heterozygous or Homozygous Familial Hypercholesterolemia Who Have Completed the Adolescent ORION-16 or ORION-13 Studies (VICTORION-PEDS-OLE)
Brief Title: Long-term Safety and Tolerability of Inclisiran in Participants With HeFH or HoFH Who Have Completed the Adolescent ORION-16 or ORION-13 Studies
Acronym: V-PEDS-OLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839C12001B; 2022-002316-23 (EudraCT Number)
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heterozygous or Homozygous Familial Hypercholesterolemia
Keywords: KJX839; heterozygous familial hypercholesterolemia; homozygous familial hypercholesterolemia; familial hypercholesterolemia; FH; inclisiran; pediatric
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — ALN-PCS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inclisiran (Experimental): Inclisiran sodium 300mg (equivalent to 284mg inclisiran*) in 1.5mL solution
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300mg (equivalent to 284mg inclisiran*) in 1.5mL solution administered subcutaneously in pre-filled syringe
  Other Names: KJX839

SUMMARY:
The purpose of this open-label, single arm, multicenter extension study is to evaluate the long-term safety and tolerability of inclisiran in participants with HeFH or HoFH who have completed the ORION-16 or ORION-13 studies.

DETAILED DESCRIPTION:
This is an open-label, single arm, multicenter study designed to evaluate long-term safety and tolerability of inclisiran. In addition, the study will provide participants the opportunity to have continued access to treatment with inclisiran.

ELIGIBILITY:
Key inclusion:

* Male and female participants with a diagnosis of HeFH or HoFH who completed the ORION-16 or ORION-13 studies
* Per investigator's clinical judgment, participant derived benefit from treatment with inclisiran in the ORION-16 or ORION-13 studies

Key exclusion:

* Participants who in the feeder inclisiran ORION-16 and ORION-13 studies either screen failed or permanently discontinued from the treatment/study for any reason or had serious safety or tolerability issues related to inclisiran treatment
* Any uncontrolled or serious disease, or any medical, physical, or surgical condition, that may either interfere with participation in the clinical study or interpretation of clinical study results, and/or put the participant at significant risk

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) | From Day 1 in the study up to the end of study visit; up to 1080 days
  Safety and tolerability: TEAEs, TESAEs (incidence, severity, relationship to study drug and discontinuation due to TEAEs)

SECONDARY OUTCOMES:
Percentage and absolute change in LDL-C from baseline in the feeder study to end of study | Baseline (of feeder study) and Day 1080
  Evaluate the long-term effect of inclisiran (from baseline of feeder study to end of study) in lowering LDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- United States (5):
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Icahn School of Med at Mt Sinai, New York, New York
  - Cincinnati Childrens Hospital MC, Cincinnati, Ohio
  - Childrens Hosp Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - Primary Childrens Medical Center, Salt Lake City, Utah
- Novartis Investigative Site, Formosa, Formosa Province, Argentina
- Brazil (2):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Québec, Quebec, Canada
- Novartis Investigative Site, Prague, Czechia
- France (2):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Freiburg im Breisgau
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Pécs, Baranya, Hungary
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Irbid, Jordan
- Novartis Investigative Site, Beirut, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Sungai Buloh, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Rotterdam, South Holland
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Russia (2):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
- Novartis Investigative Site, Poprad, Slovakia
- Novartis Investigative Site, Ljubljana, Slovenia
- South Africa (2):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Cape Town, Western Cape
- Spain (4):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Geneva, Switzerland
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Adana, Saricam
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com